CLINICAL TRIAL: NCT01784250
Title: Efficacy of Clonidine and Propranolol Versus Placebo for the Control of Anxiety During Surgical Procedures in Dentistry
Brief Title: Efficacy of Clonidine and Propranolol in Dentistry (AAA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Patricia Bermúdez Reyes, Researcher, CES University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLON000
Record Dates: First submitted 2013-01-23; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Anxiety
Keywords: Clonidine; Propranolol; Third molar; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Clonidine; Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Propanolol (Experimental): Propranolol 40mg tablets, one tablet administered 1 hour before surgery
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Placebo tablets, one tablet administered 1 hour before surgery
  Interventions: Drug: Placebo
- Clonidine (Experimental): clonidine 150mcg tablets, one tablet administered 1 hour before surgery
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine — Clonidine 150 mcg tablet single dose, to receive by mouth one hour before surgery
  Other Names: Catapresan
  Arms: Clonidine
Drug: Propranolol — Propranolol 40 mg tablet single dose, to receive by mouth one hour before surgery
  Other Names: Artensol; Inderal
  Arms: Propanolol
Drug: Placebo — Sugar pill manufactured to mimic a drug
  Arms: Placebo

SUMMARY:
The aim of the study is to determine the efficacy of clonidine and propranolol for transient anxiety management and intra and postoperative pain in patients undergoing ambulatory surgery of third molar.

DETAILED DESCRIPTION:
There will be a randomized, triple-blind, placebo-controlled clinical trial with parallel group design to determine the efficacy of the pre medication propranolol and clonidine versus placebo for reducing anxiety during third molar removal surgery. Patients will be assigned to 3 groups of 20 patients each. One group will receive 150 mcg of clonidine, the second group will receive propranolol 40mg, and the control group will receive placebo. The modified dental anxiety scale will be applied before and after surgery in order to evaluate the change in anxiety level, which will be assessed as the primary outcome. The secondary outcomes include the measurement of changes in blood pressure, heart rate and respiratory rate evaluated before, during and after surgery. Additionally, pain will be assessed through numerical pain scale at 3, 6 and 24 hours after surgery. Also, possible side effects will be identified (vomiting, nausea, dry mouth, dizziness and drowsiness). Statistical analysis: qualitative variables will be described by absolute and relative frequencies, and quantitative variables will be described by the mean along with standard deviation or the median with interquartile range depending on the distribution of the data. One-way ANOVA or Kruskal Wallis will be used (depending on the fulfillment of assumptions) in order to compare the quantitative variables amongst the groups. The chi squared test will be used to compare the qualitative variables. The confidence intervals will be estimated at 95% for all effect magnitude measurements calculated.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive patients and pre-hypertension who are undergoing elective surgery for removal of third molars.
* Age range 14 to 40 years
* Patients with dental anxiety above 13 points on the scale (MDAS).
* People who voluntarily agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* Patients receiving any medication for any chronic pathology.
* Patients of African American race, being more likely to have abnormal blood pressure.
* Patients with a history of cardiovascular disease.
* Patients with chronic systemic disease such as diabetes, hyper or hypothyroidism, Addison's syndrome, renal failure, hypertension or liver disease.
* Pregnant or breastfeeding.
* Patients diagnosed with anxiety disorder or depressive disorder

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in modified dental anxiety scale(MDAS)and vital signs (blood pressure, heart rate, respiratory rate, oxygen saturation) until four hours post treatment | (plus or minus 4 hours) after surgery

SECONDARY OUTCOMES:
Changes in Verbal Numerical Rating Scale (VNRS) at three, six, and twenty-four hours post treatment | 24 hours

OTHER OUTCOMES:
Frequency of side effects in patients treated with clonidine and propranolol compared with placebo after third molar surgery | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bermudez, Dentistry, Principal Investigator — CES University; Libia M Rodriguez, Magister, Study Director — CES University; Ana K Tamara, Physician, Principal Investigator — CES University
Locations (1):
- Cooperative University, Envigado, Antioquia, Colombia

REFERENCES:
- [Background] Ng SK, Leung WK. A community study on the relationship of dental anxiety with oral health status and oral health-related quality of life. Community Dent Oral Epidemiol. 2008 Aug;36(4):347-56. doi: 10.1111/j.1600-0528.2007.00412.x. PMID 19145721
- [Background] Kvale G, Berggren U, Milgrom P. Dental fear in adults: a meta-analysis of behavioral interventions. Community Dent Oral Epidemiol. 2004 Aug;32(4):250-64. doi: 10.1111/j.1600-0528.2004.00146.x. PMID 15239776
- [Background] Lago-Mendez L, Diniz-Freitas M, Senra-Rivera C, Seoane-Pesqueira G, Gandara-Rey JM, Garcia-Garcia A. Postoperative recovery after removal of a lower third molar: role of trait and dental anxiety. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Dec;108(6):855-60. doi: 10.1016/j.tripleo.2009.07.021. PMID 19913724
- [Background] Humphris GM, Dyer TA, Robinson PG. The modified dental anxiety scale: UK general public population norms in 2008 with further psychometrics and effects of age. BMC Oral Health. 2009 Aug 26;9:20. doi: 10.1186/1472-6831-9-20. PMID 19709436
- [Background] Hall DL, Tatakis DN, Walters JD, Rezvan E. Oral clonidine pre-treatment and diazepam/meperidine sedation. J Dent Res. 2006 Sep;85(9):854-8. doi: 10.1177/154405910608500915. PMID 16931871
- [Background] Liu HH, Milgrom P, Fiset L. Effect of a beta-adrenergic blocking agent on dental anxiety. J Dent Res. 1991 Sep;70(9):1306-8. doi: 10.1177/00220345910700091401. PMID 1918581
- [Background] Herr KA, Spratt K, Mobily PR, Richardson G. Pain intensity assessment in older adults: use of experimental pain to compare psychometric properties and usability of selected pain scales with younger adults. Clin J Pain. 2004 Jul-Aug;20(4):207-19. doi: 10.1097/00002508-200407000-00002. PMID 15218405